CLINICAL TRIAL: NCT05802043
Title: Cognitive Stimulating Interventions Improve Cognitive Self- Efficacy and Sense of Happiness Among Older Adults
Brief Title: Effect of Cognitive Stimulating Interventions on Cognitive Self-Efficacy and Sense of Happiness Among Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15012023
Record Dates: First submitted 2023-03-25; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-01

CONDITIONS: Self- Efficacy
Keywords: Sense of Happiness; Cognitive Stimulating Interventions

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Stimulating Interventions (Experimental): The study interventions will be developed by the researchers based on review of the related literature and with reference to the CST manual (Spector, et al., 2006), and review on Cognitive Stimulation (Woods et al., 2012). The study subjects of group 1, the study group, will receive the proposed interventions, the cognitive stimulation interventions through small groups of study subjects receiving 12 sessions of group activities (2 sessions/week, approximately 45- 60 minutes/session). A group size of 6 to 8 will be conducted. The interventions group will be conducted in activity rooms within the elderl club. The study subjects group 2, the control group, will receive the routine activities of the elderly club. The researchers will provide the control group with written materials related the essential cognitive stimulation interventions after ending the implementation of the proposed interventions for the study group.
  Interventions: Behavioral: Cognitive Stimulating Interventions
- Routine Club care (Active Comparator): The study subjects group 2, the control group, will receive the routine activities of the elderly club.The researchers will provide the control group with written materials related the essential cognitive stimulation interventions after ending the implementation of the proposed interventions for the study group,
  Interventions: Behavioral: Cognitive Stimulating Interventions

INTERVENTIONS:
Behavioral: Cognitive Stimulating Interventions — a quasi-experimental research design.The study subjects of group 1, the study group, will receive the proposed interventions, the cognitive stimulation interventions through small groups of study subjects receiving 12 sessions of group activities (2 sessions/week, approximately 45- 60 minutes/session). A group size of 6 to 8 will be conducted. The interventions group will be conducted in activity rooms within the elderly club.

SUMMARY:
The present study aims to determine the effect of cognitive stimulation interventions on cognitive self-efficacy and sense of happiness among older adults.

Research hypothesis:

Older adults who receive the cognitive stimulation interventions exhibit higher cognitive self-efficacy and sense of happiness than those who do not receive it.

DETAILED DESCRIPTION:
A convenient sample of eighty (80) older adults will be used according Epi info V 7.0 program calculation based on the following statistical parameters ; Population size: 250, expected frequency: 50%, confidence coefficient: 95%, acceptable error: 10%, minimum sample size = 70.

The study will include eighty (80) older adults aged 60 years and more and fulfilling the following criteria:

Inclusion criteria

1. Aged 60 years and old.
2. Able to read and write.
3. Have mild cognitive impairment: score of score of 18-23 based on the Mini Mental State Examination Scale (MMSE).
4. Have no depression: score of 0 to 4 using the Geriatric Depression Scale Short Form (GDS_SF).
5. Accept participation in the study. 6. Available at the selected setting during the time of data collection. 7. Have no pronounced impairment of their visual and auditory abilities could affect their participation in the group and make use of most of the materials in the sessions, as determined by the researchers.

The selected study subjects (80) will be randomly assigned to two equal groups of 40 older adults each as flows; Group 1, study group: include older adults who will receive the proposed interventions, cognitive stimulation interventions.

Group 2, control group: include older adults who will receive the routine activities of the elderly club.

ELIGIBILITY:
Inclusion Criteria:1. Aged 60 years and old. 2. Able to read and write. 3. Have mild cognitive impairment: score of score of 18-23 based on the Mini Mental State Examination Scale (MMSE).

4. Have no depression: score of 0 to 4 using the Geriatric Depression Scale Short Form (GDS_SF).

5. Accept participation in the study. 6. Available at the selected setting during the time of data collection.

Exclusion Criteria:

* 7. Have pronounced impairment of their visual and auditory abilities could affect their participation in the group and make use of most of the materials in the sessions, as determined by the researchers.

Ages: 60 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
I) Mini-Mental State Examination (MMS) Scale | 2 weeks
  The MMS scale was developed by Folestein et al., (1975). It used to assess cognitive function of the older adults. It contained questions concerning registration, orientation, calculation, recall, attention, and language. The MMS scale score was 30 point and classified as follows: -30. -23. -17.
  The MMS was translated into Arabic and approved to be valid and reliable (r=0.96) by El Husseini (2008). The Arabic version of this scale was used in the present study.

SECONDARY OUTCOMES:
II) Geriatric Depression Scale- Short Form (GDS-SF) | 2 weeks
  The Geriatric Depression Scale - short Form (GDS-SF), a self-report tool with 15-item developed by Yesavage et al. (1983) to assess general well-being and depression in the elderly. The older adults should select one answer either yes (1) or no (0) for their feelings over the past week. The scores ranged from 0 to 15. Items' score will be calculated for the total score. A score of 0 to 4 meant no depression, score of 5 to 8 meant mild depression, score of 9 to 11 meant moderate depression, and 12-15 meant severe depression.
  The GDS-SF was translated into Arabic and approved to be reliable (r=0.70) and valid by ElHusseini (2013). The Arabic version of this scale was used in the current study.

OTHER OUTCOMES:
III) Six -Domains Perceived Cognitive Self-Efficacy for Older Adults Structured Interview Questionnaire | 2 weeks
  This tool will be developed by the researchers to assess the cognitive self-efficacy among older adults. It composed of 40 items related to six domains covering six cognitive functions (Everyday Memory, Language, Visuospatial Abilities, Planning, Organization, and Divided attention). Each domain contains several cognitive task related to this domain. Older adults asked to rate how certain they are that they can do each cognitive task. They rate the degree of confidence in their cognitive abitity by recording a number from 0 to 10, next to each statement, where 0 means cannot do at all, 5 moderately certain can do, and 10 indicates highly certain can do.the total score ranges from 0 to 400. The higher the score is the higher cognitive self-efficacy.
IV) The Subjective Happiness Scale (SHS): | 2 weeks
  The Subjective Happiness Scale is a 4-item scale that developed by Lyubomirsky, et al., (1999) to measure subjective happiness. Each item is completed by choosing one of 7 options that finish a given sentence fragment. The options are different for each of the four questions. Two items ask respondents to characterize themselves using both absolute ratings and ratings relative to peers, whereas the other two items offer brief descriptions of happy and unhappy individuals and ask respondents the extent to which each characterization describes them. The average of the item scores is an overall measure sense of happiness with high scores indicating greater sense of happiness.

CONTACTS AND LOCATIONS:
Overall Officials: Eman Taha, professor, Study Chair — Egypt Faculty of Nursing Alexandria, Egypt
Locations (1):
- Faculty of Nursing, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Apostolo J, Bobrowicz-Campos E, Holland C, Cano A. One small step in frailty research, a giant leap in evidence based practice. JBI Database System Rev Implement Rep. 2018 Jan;16(1):1-3. doi: 10.11124/JBISRIR-2017-003672. No abstract available. PMID 29324548
- [Background] Coen RF, Flynn B, Rigney E, O'Connor E, Fitzgerald L, Murray C, Dunleavy C, McDonald M, Delaney D, Merriman N, Edgeworth J. Efficacy of a cognitive stimulation therapy programme for people with dementia. Ir J Psychol Med. 2011 Sep;28(3):145-147. doi: 10.1017/S0790966700012131. PMID 30200025
- [Background] Feng L, Zin Nyunt MS, Gao Q, Feng L, Yap KB, Ng TP. Cognitive Frailty and Adverse Health Outcomes: Findings From the Singapore Longitudinal Ageing Studies (SLAS). J Am Med Dir Assoc. 2017 Mar 1;18(3):252-258. doi: 10.1016/j.jamda.2016.09.015. Epub 2016 Nov 9. PMID 27838339
- [Background] Kelly ME, Finan S, Lawless M, Scully N, Fitzpatrick J, Quigley M, Tyrrell F, O'Regan A, Devane A. An evaluation of community-based cognitive stimulation therapy: a pilot study with an Irish population of people with dementia. Ir J Psychol Med. 2017 Sep;34(3):157-167. doi: 10.1017/ipm.2016.23. PMID 30115146